CLINICAL TRIAL: NCT03348852
Title: Assoziation Zwischen Funktionellen Gehirnveränderungen Und Der Schmerzwahrnehmung Bei Patienten Mit Chronisch entzündlicher Darmerkrankung Mittels fMRT
Brief Title: Association Between Functional Changes in the Brain and the Perception of Pain in Patients With Inflammatory Bowel Diseases (IBD) - Measured With Functional Magnetic Resonance Imaging.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Magdalena S. Prüß née Volz, Dr. med. Magdalena Sarah Prüß (geb. Volz), Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA4/017/16
Record Dates: First submitted 2017-05-22; First posted 2017-11-21 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Active transcranial direct current stimulation
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Sham transcranial direct current stimulation
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Device: Transcranial direct current stimulation Transcranial direct current stimulation over the motor cortex.
  Other Names: tDCS

SUMMARY:
In the study the investigators aim to test whether transcranial direct current stimulation (tDCS)-induced pain reduction is in association with functional changes in the brain measured with functional magnetic resonance imaging (fMRI) in patients with chronic inflammatory bowel diseases (IBD).

Hypothesis: Transcranial direct current stimulation can reduce the perception of pain in patients with chronic inflammatory bowel diseases, which is in association with changes in the brain measured via fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease
* Chronic pain (more than 3 months)
* Pain (VAS > 3/10)

Exclusion Criteria:

* Contraindication to transcranial direct current stimulation
* Contraindications to functional magnetic resonance imaging (fMRI)
* Pregnancy
* Sever internal or psychiatric condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-01-24 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional and/or structural changes in the brain measured with cerebral MRI | 2 week
  Participants will be followed for 2 weeks
Changes in pain measured with visual analogue scale | 2 weeks
  Participants will be followed for 2 weeks
Changes in perception of pain measured with an algometer (pain pressure threshold) | 2 weeks
  Participants will be followed for 2 weeks

SECONDARY OUTCOMES:
Changes in questionnaire "quality of life" | 2 weeks
  questionnaire
Changes in functional symptoms | 2 weeks
  Questionnarie: irritable bowel syndrome - severity scoring system (IBS-SSS)
Changes in activity indices | 2 weeks
  Harvey-Bradshaw Index (HBI) or simple clinical colitis activity index
Changes in pain catastophizing scale | 2 weeks
Changes in inflammation biomarker (blood - C-reactive protein) | 2 weeks
Changes in inflammation biomarker (stool - calprotectin) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena S Prüß-Volz, MD, Principal Investigator — Charite University
Locations (1):
- Charité University Medicine, Berlin, Germany